CLINICAL TRIAL: NCT00983151
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study to Evaluate the Efficacy and Safety of Two Doses of Tramadol Hydrochloride Orally Disintegrating Tablets in Male Subjects With Premature Ejaculation
Brief Title: Study to Evaluate Efficacy and Safety in Males Subjects With Premature Ejaculation
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: BVF-324-301
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2012-08-27 (Estimated); Status verified 2010-10

CONDITIONS: Premature Ejaculation
MeSH Terms: conditions — Premature Ejaculation | interventions — Tramadol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental)
  Interventions: Drug: Tramadol Hydrochloride & Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Tramadol Hydrochloride & Placebo

INTERVENTIONS:
Drug: Tramadol Hydrochloride & Placebo — 89 mg or a lesser dose of 62 mg if side effects are experienced one tablet at least two hours before sexual intercourse (maximum of one tablet every 20 hours) Subject will take the study drug for about 27 weeks

SUMMARY:
The purpose of this clinical trial is to test an experimental drug therapy called Tramadol Hydrochloride (HCl) Orally Disintegrating Tablets (ODT) ("Tramadol HCl ODT" or the "study drug"). The subject and his partner are being asked to be in this clinical trial because they have a condition called premature ejaculation.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible for study participation if all of the following criteria are met:

1. Male subject and female partner to provide written informed consent prior to the performance of any study-specific procedures;
2. Candidates will be male subjects aged 18-65 years inclusive, with lifelong premature ejaculation ("lifelong" is defined as starting at the time the subject became sexually active) with an IELT of ≤120 seconds as documented at Visit 2.
3. History of premature or rapid ejaculation, determined by following criteria in the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM IV TR):

   1. Persistent or recurrent ejaculation with minimal sexual stimulation before, on, or shortly after vaginal insertion and before the person wishes it, taking into account factors that affect duration of the excitement phase such as age, novelty of the sexual partner or situation and recent frequency of sexual activity
   2. The disturbance causes marked distress or interpersonal difficulty
   3. The premature ejaculation is not due exclusively to the direct effects of a substance (ab)use
4. In a stable, monogamous, heterosexual relationship (> 6 months).
5. Willing and able to take study medication as directed at least 2 hours prior to sexual intercourse according to protocol;
6. Subject willing and able to complete the therapeutic trial, all sexual behavior logs, IELT assessments, questionnaires and interviews:
7. Female sexual partner willing and able to complete the therapeutic trial, all sexual behavior logs, IELT assessments, questionnaires and interviews;
8. Able to understand the study procedures, complete the assessments, and communicate with study personnel;
9. Subject and partner willing and able to engage in vaginal intercourse at least three times between visits to yield at least three events of vaginal intercourse ;
10. Subject and partner willing to use a reliable contraceptive method during the trial period if the partner is not menopausal;
11. Partner willing to take pregnancy tests at Visits 1 and 2
12. Subject willing to list and document prescription and non-prescription drug use during the study;
13. Have a negative urine drug screen at Visits 1 and 2;
14. Be in good general health as determined by medical history and physical examination and expected by the Investigator to complete the study as designed.

Exclusion Criteria:

Subjects are not eligible for study participation if any of the following criteria are met:

1. Premature ejaculation attributable to situational or relationship issues;
2. Evidence or a history of other significant psychiatric disorder as defined as requiring therapy or medication;
3. Subjects who in the Investigator's opinion are at significant risk of suicide.
4. Physical illnesses i.History of seizures ii.Prostatitis (current) iii.Urethritis or other urinary tract infections (current) iv.Prior genital surgery (other than vasectomy or circumcision) v.Uncontrolled Diabetes mellitus vi.Respiratory Depression vii.Thyroid disease viii.Chronic moderate to severe neurological disease ix.Significant heart disease treated with cardiac drugs x.Chronic liver disease xi.Chronic kidney disease xii.History of cardiovascular disease (myocardial infarction, congestive heart failure, angina, coronary artery disease or stroke) xiii.Known to be a carrier of the hepatitis B surface antigen, hepatitis C virus antibody, and/or immunodeficiency virus-1 and/ or 2 antibodies xiv.Other disorder that may cause sexual dysfunction
5. Other sexual dysfunction:

   i.Erectile dysfunction. As defined by the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM IV TR), the diagnostic criteria for male erectile disorder (302,72) erectile dysfunction includes:

   A.Persistent or recurrent inability to attain, or to maintain until completion of the sexual activity, an adequate erection.

   B.The disturbance causes marked distress or interpersonal difficulty. ii.Primary reduced sexual desire unrelated to premature ejaculation
6. Sexual intercourse usually less than once per week;
7. Partner sexual dysfunction (for example dyspareunia or other conditions considered relevant);
8. Current use of dapoxetine;
9. Current use of any tramadol;
10. Sensitivity to phenylketone;
11. Any history of abuse of prescription opioids and/or illicit/illegal addictive drugs;
12. Has a known hypersensitivity to heparin or history of heparin induced thrombocytopenia;
13. Use of medication, within the preceding 30 days, with potential to cause sexual dysfunction: (See Appendix 2 for a list of excluded medications) i.Antidepressants - all types

    ii.Antipsychotic medication

    iii.Antihypertensive medication, unless on a stable dose > 6 months

    iv.Hormonal drugs

    v.Chemotherapy

    vi.Others: cimetidine, clofibrate,quinidine
14. Recent psychotropic drug use (within the past 30 days);
15. A history of alcohol abuse or dependence within the past 6 months as defined by the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM IV TR);
16. Initiation of psychosexual counseling during the screening, baseline or treatment periods;
17. Partner positive pregnancy test at Visit 1 or 2;
18. History of clinically significant intolerance or a known hypersensitivity to tramadol, such that treatment with it is contraindicated;
19. The Investigator anticipates that the subject will be unable to comply with the protocol;
20. Received any investigational drug within 30 days prior to Visit 1 or is scheduled to receive an investigational drug during the course of this study;
21. Has preplanned surgery or procedures that would interfere with the course of the study.
22. A family member (other than the female partner), a staff member, or relative of a staff member..
23. Significant laboratory abnormality as determined by the Investigator at Visit 1;
24. Significant ECG abnormality at Visit 1 as determined by the Investigator;
25. Any other illnesses, conditions or practices that in the Investigator's opinion could interfere with the collection and/or interpretation of study results (couples using the "Withdrawal Method" of birth control will be excluded from the study).

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Increase in IELT (Intravaginal ejaculatory time) | Per attempt at sexual intercourse

SECONDARY OUTCOMES:
Efficacy of using Tramadol for Premature Ejaculation. | At each attempt

CONTACTS AND LOCATIONS:
Overall Officials: Hubert Claes, MD, Principal Investigator — Clinique St Jean
Locations (38):
- Innsbruck Medical university, Innsbruck, Austria
- Belgium (6):
  - Ziekenhuisnelwerk Antwerpen (ZNA), Campus Stuvenberg-St. Erasmus, Antwerp
  - Clinique St. Jean, Depart. of Urology, Blvd du Jardin Botanique, 32, Brussels
  - UZ Brussel, Laarbeeklaan 101, Brussels
  - Universitair Ziekenhuls Antwerpen (UZA), Wirjkstraat 10, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - CHU Sart Tilman, Liège
- France (12):
  - CHU de Nimes-Groupe Hospitalo-Universitaire, Pharmacie Secteur Essals Cliniques,, Cedex
  - Hopital Raymond Poincar'e, 104 Bvld. Raymond Poincar'e, Garches
  - Hopital Henry Gabrielle, Laval
  - CETPARPjj, Lille
  - hopital Edouard Herriot, Lyon
  - Institut de Medecine Sexuelle, Marseille
  - Hopital Pasteur, Nice
  - Porle Bouqueyre, Parc Saint-Maur
  - 11 rue Magellan, Paris
  - Cabinet medical, Paris
  - 76 rue d'Antain, 35700 Rennes, Rennes
  - Cabinet medical, 10 rue de la Trinite, Toulouse
- Germany (6):
  - Dederweg 2-4, Frankfurt
  - University Hospital Halle, Halle
  - Institut fur Mannergesundheit Universitakslinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover Zentrum for Seelische Gesundhelt, Hanover
  - Abetellung for Andrologie & Urologie PAN-Kilnik am Neumarkt, Koin
  - PUR/R Praxisklinik Urologie 3 Rhein Ruhr, Mühlheim
- Netherlands (2):
  - Academic Medical Center, Depart. of Urology, Amsterdam
  - Geert Grooteplein Zuid, Nijmegen
- Spain (4):
  - Hospital Universitario Reina Sofla, Córdoba
  - Hospital Universitario Fundacion Alcordon, Madrid
  - Clinica El Angel, Málaga
  - Hospital Universitario Virgen de Rocio, Seville
- Sweden (7):
  - DW Medical, Eskilstuna
  - Carlanderska Sjukhuset, Gothenburg
  - Urohalsan, Jönköping
  - ProbarE AB, Lund
  - ProbarE AB, Solna
  - Karolinska University hospital-Huddinge, Stockholm
  - S3 Clinical Research Centers, Vällingby

REFERENCES:
- [Derived] Bar-Or D, Salottolo KM, Orlando A, Winkler JV; Tramadol ODT Study Group. A randomized double-blind, placebo-controlled multicenter study to evaluate the efficacy and safety of two doses of the tramadol orally disintegrating tablet for the treatment of premature ejaculation within less than 2 minutes. Eur Urol. 2012 Apr;61(4):736-43. doi: 10.1016/j.eururo.2011.08.039. Epub 2011 Aug 30. PMID 21889833